CLINICAL TRIAL: NCT00648206
Title: Retrospective Study of Unrequested Analytical Data in DUID-cases From a 2 Week Period
Brief Title: Testing Alcohol Only Samples for Drugs and Drugs Only Samples for Alcohol
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Ministry of Internal Affairs, Finland (Unknown); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: KTL 419-9
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Driving Under the Influence
Keywords: driving under the influence; psychoactive substances; blood samples; Prevalence of psychoactive substances in road traffic
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Observational Model: Case-Crossover
Biospecimen Retention: Samples With DNA — Whole blood samples are collected for the study. However no DNA detection is done at any point in the study. The laboratory where the samples are analysed does not analyse DNA. DNA is not relevant for this study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: drivers of motorised vehicles suspected of driving under the influence of psychoactive drugs or alcohol
- 2: drivers stopped in police traffic controls and breathalysed positive for alcohol

SUMMARY:
This study intends to supply information about the prevalence of psychoactive drugs and alcohol in suspected DUI samples which are suspected of only one of these rather than both drugs and alcohol.

Police samples for suspected DUI samples that have been sent for alcohol analysis or drug analysis only will be screened for drugs and alcohol respectively.

DETAILED DESCRIPTION:
There are 3 different possibilities for forensic analysis of suspected driving under the influence samples. Testing for alcohol or drugs only or testing for both alcohol and drugs.

Often if the primary suspicion of the apprehending police officer is of driving under the influence of drugs or alcohol then only laboratory analysis concerning that primary suspicion is requested.

The study aims to provide information about those 'missed cases' where only analysis for drugs or alcohol is carried out. Traffic police samples from a 2 week period are to be screened for both drugs and alcohol, even if the primary suspicion is only one of these.

The study is part of the EU-project DRUID. Altogether 13 European countries are participating in DRUID.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* driver of a motorised vehicle

Exclusion Criteria:

* 17 years or younger
* not the driver of a motorised vehicle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: drivers of motorised vehicles in general road traffic
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
assessment of both alcohol and drugs in suspected DUI cases | 2 weeks

SECONDARY OUTCOMES:
prevalence of psychoactive substances in the general driving population | three years

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Lillsunde, Dr, Principal Investigator — National Public Health Institute, Helsinki, Finland
Locations (1):
- National Public Health Institute, Helsinki, Finland

REFERENCES:
- See also: Official home page of the EU-project — http://www.druid-project.eu